CLINICAL TRIAL: NCT02042131
Title: Brief Interventions for Short-Term Suicide Risk Reduction in Military Populations
Acronym: BISSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Craig Bryan, PI, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01481; W81XWH-10-2-0181 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Suicide; Suicidal Ideation
Keywords: suicide; suicidal ideation; ambivalence; suicide ambivalence; reasons for living; reasons for dying; military; veteran; clinical trial; cognitive behavioral therapy; psychotherapy; crisis; Treatment As Usual (TAU); Crisis Response Plan (CRP); Enhanced Crisis Response Plan (E-CRP)
MeSH Terms: conditions — Suicide; Suicidal Ideation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment As Usual (TAU) (Active Comparator): TAU includes the following intervention components:
  1. suicide risk assessment
  2. supportive listening
  3. provision of professional and crisis contact information
  4. referral to mental health treatment and community resources
  5. verbal contract for safety
  Interventions: Behavioral: Treatment As Usual (TAU)
- Standard Crisis Response Plan (S-CRP) (Experimental): CRP includes the following intervention components:
  1. suicide risk assessment
  2. supportive listening
  3. identify personal warning signs
  4. identify self-management skills
  5. identify social support contacts
  6. provision of professional and crisis contact information
  7. referral to mental health treatment and community resources
  Interventions: Behavioral: Standard Crisis Response Plan (S-CRP); Behavioral: Enhanced Crisis Response Plan (E-CRP)
- Enhanced Crisis Response Plan (E-CRP) (Experimental): The E-CRP includes the following intervention components:
  1. suicide risk assessment
  2. supportive listening
  3. identify personal warning signs
  4. identify self-management skills
  5. identify reasons for living
  6. identify social support contacts
  7. provision of professional and crisis contact information
  8. referral to mental health treatment and community resources
  Interventions: Behavioral: Enhanced Crisis Response Plan (E-CRP)

INTERVENTIONS:
Behavioral: Treatment As Usual (TAU)
  Other Names: Usual Care; Enhanced Care; Enhanced Care As Usual
  Arms: Treatment As Usual (TAU)
Behavioral: Standard Crisis Response Plan (S-CRP)
  Other Names: Safety Plan
  Arms: Standard Crisis Response Plan (S-CRP)
Behavioral: Enhanced Crisis Response Plan (E-CRP)
  Other Names: Safety Plan
  Arms: Enhanced Crisis Response Plan (E-CRP); Standard Crisis Response Plan (S-CRP)

SUMMARY:
The purpose of the proposed study is to identify the most effective brief interventions for reducing short-term risk for suicide attempts in "real world" military triage settings, and to identify potential mechanisms of change underlying the interventions' impact on subsequent suicide attempts. We will randomize 360 patients to one of three commonly-used crisis interventions delivered as routine care in the mental health triage system: (1) Treatment As Usual (TAU); (2) Standard Crisis Response Plan (S-CRP); or (3) Enhanced Crisis Response Plan with Reasons For Living (E-CRP). The following hypotheses will be tested:

1. The enhanced crisis response plan (E-CRP) intervention will contribute to significantly decreased risk for suicide attempts and hospitalization during follow-up relative to the standard crisis response plan alone (S-CRP) and treatment as usual (TAU).
2. The standard crisis response plan (S-CRP) intervention will contribute to significantly decreased risk for suicide attempts and hospitalization during follow-up relative to treatment as usual (TAU).
3. Greater ambivalence about suicide and faster recall of reasons for living will mediate the relationship between intervention and reduced risk for suicide attempt during follow-up.

DETAILED DESCRIPTION:
The CRP has been proposed as an alternative to TAU for the short-term management of suicidal patients and is now in widespread use, but has never been empirically tested. The CRP is purported to reduce suicide risk via unique mechanisms that directly suicide risk, notably suicidal ambivalence (i.e., the relative balance between the wish to live and the wish to die) and problem solving. Because suicidal ambivalence has gained support as an active mechanism for reducing suicide risk, the present study will also seek to augment this underlying mechanism by directly engaging the suicidal patient in a discussion about their reasons for living, thereby potentially increasing the potency of the CRP.

The present study therefore entails a component analysis of crisis interventions. As such, we anticipate ordered effects, whereby the S-CRP and E-CRP conditions will show significantly better outcomes than TAU, and E-CRP will demonstrate significantly better outcomes than the standard CRP condition.

ELIGIBILITY:
Inclusion Criteria:

* Active duty
* 18 years of age or older
* Reporting current suicidal ideation with intent to die, or a suicide attempt within the past two weeks
* Able to speak and understand the English language
* Able to complete the informed consent process

Exclusion Criteria:

* Severe psychiatric or medical conditions that preclude the ability to provide informed consent or participation in outpatient treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig J Bryan, PsyD, ABPP, Principal Investigator — National Center for Veterans Studies & The University of Utah; Tracy A Clemans, PsyD, Study Director — National Center for Veterans Studies & The University of Utah
Locations (1):
- Fort Carson, Colorado Springs, Colorado, United States

REFERENCES:
- [Derived] Bryan CJ, Mintz J, Clemans TA, Burch TS, Leeson B, Williams S, Rudd MD. Effect of Crisis Response Planning on Patient Mood and Clinician Decision Making: A Clinical Trial With Suicidal U.S. Soldiers. Psychiatr Serv. 2018 Jan 1;69(1):108-111. doi: 10.1176/appi.ps.201700157. Epub 2017 Oct 2. PMID 28967323
- [Derived] Lowder EM, Rade CB, Desmarais SL. Effectiveness of Mental Health Courts in Reducing Recidivism: A Meta-Analysis. Psychiatr Serv. 2018 Jan 1;69(1):15-22. doi: 10.1176/appi.ps.201700107. Epub 2017 Aug 15. PMID 28806894
- See also: National Center for Veterans Studies — http://veterans.utah.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment As Usual (TAU): TAU includes the following intervention components:
  1. suicide risk assessment
  2. supportive listening
  3. provision of professional and crisis contact information
  4. referral to mental health treatment and community resources
  5. verbal contract for safety
  Treatment As Usual (TAU)
- Standard Crisis Response Plan (S-CRP): CRP includes the following intervention components:
  1. suicide risk assessment
  2. supportive listening
  3. identify personal warning signs
  4. identify self-management skills
  5. identify social support contacts
  6. provision of professional and crisis contact information
  7. referral to mental health treatment and community resources
  Treatment As Usual (TAU)
  Crisis Response Plan (CRP)
- Enhanced Crisis Response Plan (E-CRP): The E-CRP includes the following intervention components:
  1. suicide risk assessment
  2. supportive listening
  3. identify personal warning signs
  4. identify self-management skills
  5. identify reasons for living
  6. identify social support contacts
  7. provision of professional and crisis contact information
  8. referral to mental health treatment and community resources
  Treatment As Usual (TAU)
  Crisis Response Plan (CRP)
  Enhanced Crisis Response Plan (E-CRP)
Period: Overall Study
Arm/Group | Treatment As Usual (TAU) | Standard Crisis Response Plan (S-CRP) | Enhanced Crisis Response Plan (E-CRP)
Started | 32 | 32 | 33
Completed | 32 | 32 | 33
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment As Usual (TAU) | Standard Crisis Response Plan (S-CRP) | Enhanced Crisis Response Plan (E-CRP) | Total
Number analyzed (Participants) | 32 | 32 | 33 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (5.3) | 27.0 (6.9) | 26.0 (6.8) | 26.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 5 | 21
  Male | 24 | 24 | 28 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 7
  Not Hispanic or Latino | 30 | 30 | 30 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Black or African American | 5 | 7 | 3 | 15
  White | 23 | 19 | 23 | 65
  More than one race | 2 | 3 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Estimated Proportion of Participants With Suicide Attempt
Description: Suicide attempts were assessed using the Suicide Attempt Self Injury Interview (SASII; Linehan et al., 2006). The SASII is a valid and reliable clinician-administered interview for categorizing suicide-related and self-injurious behaviors. Suicide attempt was defined as behavior that is self-directed and deliberately results in injury or the potential for injury to oneself for which there is evidence, whether implicit or explicit, of suicidal intent
Time Frame: 6 months
Population: all participants enrolled, regardless of dropout or withdrawal
Measure: Number; unit: estimated proportion of participants
Groups:
- Standard Crisis Response Plan (S-CRP): CRP includes the following intervention components:
  1. suicide risk assessment
  2. supportive listening
  3. identify personal warning signs
  4. identify self-management skills
  5. identify social support contacts
  6. provision of professional and crisis contact information
  7. referral to mental health treatment and community resources
  Standard Crisis Response Plan (S-CRP)
  Enhanced Crisis Response Plan (E-CRP)
- Enhanced Crisis Response Plan (E-CRP): The E-CRP includes the following intervention components:
  1. suicide risk assessment
  2. supportive listening
  3. identify personal warning signs
  4. identify self-management skills
  5. identify reasons for living
  6. identify social support contacts
  7. provision of professional and crisis contact information
  8. referral to mental health treatment and community resources
  Enhanced Crisis Response Plan (E-CRP)
Arm/Group | Treatment As Usual (TAU) | Standard Crisis Response Plan (S-CRP) | Enhanced Crisis Response Plan (E-CRP)
Number analyzed (Participants) | 32 | 32 | 33
estimated proportion of participants | 0.19 | 0.03 | 0.06
Statistical Analysis 1: Comparison: Treatment As Usual (TAU) vs Standard Crisis Response Plan (S-CRP) vs Enhanced Crisis Response Plan (E-CRP); Omnibus test of all three groups; Test type: Superiority; p = .082, Log Rank
Statistical Analysis 2: Comparison: Treatment As Usual (TAU) vs Standard Crisis Response Plan (S-CRP) vs Enhanced Crisis Response Plan (E-CRP); Planned contrast #1: TAU vs. S-CRP/E-CRP; Test type: Superiority; p = .028, Log Rank
Statistical Analysis 3: Comparison: Treatment As Usual (TAU) vs Standard Crisis Response Plan (S-CRP) vs Enhanced Crisis Response Plan (E-CRP); Planned contrast #1: TAU vs. S-CRP/E-CRP; Test type: Superiority; p = .040, Regression, Cox; Cox Proportional Hazard = 0.24, 95% CI 2-sided [0.06 to 0.96]

2. Secondary Outcome: Beck Scale for Suicide Ideation (BSSI)
Description: The BSSI is used to evaluate the intensity of the patient's specific attitudes, behaviors, and plans to make a suicide attempt. BSSI total score was used as the outcome measure. Total scores range from 0 to 38, with higher scores indicating more severe suicide ideation.
Time Frame: 1 month, 3 months, and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Standard Crisis Response Plan (S-CRP): CRP includes the following intervention components:
  1. suicide risk assessment
  2. supportive listening
  3. identify personal warning signs
  4. identify self-management skills
  5. identify social support contacts
  6. provision of professional and crisis contact information
  7. referral to mental health treatment and community resources
  Treatment As Usual (TAU)
  Crisis Response Plan (S-CRP)
- Enhanced Crisis Response Plan (E-CRP): The E-CRP includes the following intervention components:
  1. suicide risk assessment
  2. supportive listening
  3. identify personal warning signs
  4. identify self-management skills
  5. identify reasons for living
  6. identify social support contacts
  7. provision of professional and crisis contact information
  8. referral to mental health treatment and community resources
  Treatment As Usual (TAU)
  Crisis Response Plan (S-CRP)
  Enhanced Crisis Response Plan (E-CRP)
Arm/Group | Treatment As Usual (TAU) | Standard Crisis Response Plan (S-CRP) | Enhanced Crisis Response Plan (E-CRP)
Number analyzed (Participants) | 32 | 32 | 33
units on a scale
  1 month | 8.4 (1.4) | 5.3 (1.4) | 3.5 (1.5)
  3 months | 5.8 (1.5) | 6.0 (1.5) | 3.3 (1.6)
  6 months | 7.3 (1.5) | 2.5 (1.6) | 1.9 (1.5)
Statistical Analysis 1: Comparison: Treatment As Usual (TAU) vs Standard Crisis Response Plan (S-CRP) vs Enhanced Crisis Response Plan (E-CRP); Omnibus test comparing all three groups; Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Treatment As Usual (TAU) vs Standard Crisis Response Plan (S-CRP) vs Enhanced Crisis Response Plan (E-CRP); Planned contrast #1: TAU vs. S-CRP/E-CRP; Test type: Superiority; p < 0.001, Mixed Models Analysis

3. Secondary Outcome: Inpatient Psychiatric Hospitalization Days
Description: Mean number of days of inpatient psychiatric hospitalization
Time Frame: 6 months
Measure: Mean (Standard Error); unit: days
Arm/Group | Treatment As Usual (TAU) | Standard Crisis Response Plan (S-CRP) | Enhanced Crisis Response Plan (E-CRP)
Number analyzed (Participants) | 32 | 32 | 33
days | 2.5 (0.6) | 0.9 (0.2) | 1.2 (0.3)
Statistical Analysis 1: Comparison: Treatment As Usual (TAU) vs Standard Crisis Response Plan (S-CRP) vs Enhanced Crisis Response Plan (E-CRP); Planned contrast #1: TAU vs. S-CRP/E-CRP; Test type: Superiority; p < 0.001, Mixed Models Analysis

4. Other Pre Specified Outcome: Number of Participants Who Were Admitted for Psychiatric Hospitalization Immediately Post-intervention by a Blinded Clinician
Description: Doctoral-level clinicians (i.e., physicians or psychologists) who were blind to treatment condition made a determination regarding psychiatric inpatient admission (either admit or not admit) immediately following the intervention.
Time Frame: Immediately post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual (TAU) | Standard Crisis Response Plan (S-CRP) | Enhanced Crisis Response Plan (E-CRP)
Number analyzed (Participants) | 32 | 32 | 33
Participants | 6 | 5 | 1
Statistical Analysis 1: Comparison: Treatment As Usual (TAU) vs Standard Crisis Response Plan (S-CRP) vs Enhanced Crisis Response Plan (E-CRP); Omnibus test of all groups; Test type: Superiority; p = 0.040, Chi-squared
Statistical Analysis 2: Comparison: Treatment As Usual (TAU) vs Standard Crisis Response Plan (S-CRP) vs Enhanced Crisis Response Plan (E-CRP); Planned contrast #2: E-CRP vs. TAU/S-CRP; Test type: Superiority; p = 0.045, Chi-squared; Odds Ratio (OR) = 0.1, 95% CI 2-sided [0.002 to 0.9]

ADVERSE EVENTS:
Arm/Group | Treatment As Usual (TAU) | Standard Crisis Response Plan (S-CRP) | Enhanced Crisis Response Plan (E-CRP)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 1/33
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 1/33
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment As Usual (TAU) (N=32) | Standard Crisis Response Plan (S-CRP) (N=32) | Enhanced Crisis Response Plan (E-CRP) (N=33)
Death by suicide (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Staffing changes at the research site resulted in a one year suspension of recruitment by the IRB and the inability to meet planned recruitment goals. In all, 97 participants were enrolled, approximately one-quarter of the original goal (N=360).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No